CLINICAL TRIAL: NCT01210586
Title: Tobacco Cessation in Postmenopausal Women - Part I & Part II
Brief Title: Tobacco Cessation in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2002NT050
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: HRT; Non-HRT; Continued Smoking; Smoking Abstinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine Patch (Active Comparator): Nicotine Patch for Smoking Cessation
  Interventions: Behavioral: Part 2
- Placebo Patch (Placebo Comparator)
  Interventions: Behavioral: Part 2

INTERVENTIONS:
Behavioral: Part 2 — Comparing smoking symptomatology by HRT and nicotine patch status using a 2x2 randomized design.

SUMMARY:
This study investigated whether being on transdermal hormone replacement therapy (HRT) influenced smoking cessation variables in postmenopausal women undergoing short-term abstinence from cigarettes. Women were recruited into two groups according to their pre-enrollment medication status - currently on HRT (n = 17) or not on HRT (n = 13). The HRT group had their prior medication replaced with a standard 0.1 mg estradiol transdermal system and 2.5 mg of Cycrin daily. Following two weeks of medication adjustment, participants continued smoking as usual for one week, at which time baseline measurements were taken. For the remaining two weeks, participants were instructed to quit smoking. They were provided with smoking cessation counseling and monitored for abstinence. Data were collected during five clinic visits on all dependent measures: Minnesota Nicotine Withdrawal Scale, Beck Depression Inventory (BDI) Scale, Profile of Mood States, Motor Speed Tasks, and Reaction Time Test.

Part II is identical to Part I, except it randomizes participants to use nicotine patch or not.

ELIGIBILITY:
Inclusion Criteria:

* 40-79 years old
* Clinical Menopause
* > 15 cigarettes per day for at least one year
* Experienced nicotine withdrawal based on DSM IV

Exclusion Criteria:

* Currently obtaining nicotine from other sources
* Abnormal vaginal bleeding
* unstable health
* history of stroke or embolism
* history of abnormal thyroid function
* significant skin disorders
* active psychiatric disease

Ages: 40 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 1999-01; Primary Completion 2004-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
During short term smoking abstinence, do the beneficial effects of nicotine replacement therapy on acute symptomatology differ in women who use and do not use hormone replacement therapy? | Outcome was measured after 1 baseline week and a 2 week quit

CONTACTS AND LOCATIONS:
Overall Officials: Sharon S Allen, MD, PhD, Principal Investigator — University of Minnesota